CLINICAL TRIAL: NCT00414115
Title: Canadian Pharmacogenomics Network for Drug Safety
Brief Title: National Active Surveillance Network and Pharmacogenomics of Adverse Drug Reactions in Children
Status: Recruiting | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: Genome Canada (Other); Genome British Columbia (Industry); Child and Family Research Institute (Other); Western University, Canada (Other); Provincial Health Services Authority British Columbia (Other); Health Canada (Other Government); Canada Gene Cure (Unknown); Eli Lilly and Company (Industry); Pfizer (Industry); Merck Sharp & Dohme LLC (Industry); Canadian Society of Clinical Pharmacology (Unknown); Canadian Institutes of Health Research (CIHR) (Other Government); Canada Foundation for Innovation (Other); British Columbia Clinical Genomics Network (Other)
Responsible Party: Principal Investigator, Bruce Carleton, Study Principal Investigator, University of British Columbia
Other Study IDs: H04-70358; CW Health Centre of BC; W04-0138
Record Dates: First submitted 2006-12-19; First posted 2006-12-21 (Estimated); Last update posted 2025-03-27 (Actual); Status verified 2024-05

CONDITIONS: Adverse Drug Reaction (ADR)
Keywords: Observational controlled study; Genomic biomarkers; Adverse drug reaction; In children OR adults
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is (1) to identify and collect samples from children and adults who take drugs and have adverse drug reactions AND children and adults who take drugs and do not experience any adverse drug effects; (2) to determine if genetic differences between the two groups contribute to causing the adverse drug reactions; and (3) to develop patient specific drug dosing guidelines to prevent future adverse drug reactions. We also wish to compare the use of prescription drugs, medical and hospital services and vital statistics between BC participants who experience adverse drug reactions and those who do not.

Study hypothesis: Genetic differences may contribute to patients' response to drugs and may be responsible for adverse drug reactions.

DETAILED DESCRIPTION:
CPNDS will identify ADR predictive markers by comparing DNA and plasma samples from patients that suffer ADRs with samples from control populations that are stratified by medication type and age. The GATC will obtain its clinical material for ADR patients mainly, from hospital-based active surveillance network across Canada's major hospitals.

1. CPNDS will examine known SNPs in candidate genes related to the ADR (i.e. drug metabolism genes, drug transporter genes, drug target genes, and other disease-specific genes or genes related to the physiological pathway of the ADR.) 2. CPNDS will discover novel ADR predictive SNPs and mutations by sequencing DNA samples from our patient cohorts. CPNDS will also genotype and sequence DNA samples from populations of controls that received the same drugs, but did not suffer ADRs; and a second population of control patients who represent a random sample of the population of known ethnic backgrounds.

Novel ADR predictive SNPs and mutations will be functionally validated by pharmacokinetic approaches applied to time course analysis of drug concentrations for each specific genotype. Pharmacokinetic studies will also be used to determine the drug concentration in patients to characterize possible mechanisms of the ADR, translating into rational approaches to the choice of candidate genes to be examined in the genomic analyses.

The cost-effectiveness of an ADR screening program for the prevention of ADRs in children and adults will be calculated in detailed health-economic studies.

ELIGIBILITY:
Inclusion Criteria:

* Children under 19 years who have taken drugs.
* Biological parents of children who have had an ADR.
* Patients/parents who speak and understand English (except in Quebec).
* Adults (for validation of findings in children)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Children under 19 years who have taken drugs and adults to replicate findings in children
Sampling Method: Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2005-08; Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Determine the role of genetic and clinical factors in adverse drug reactions to develop risk mitigation strategies. | December 2018

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Carleton, Pharm. D., Principal Investigator — University of British Columbia; Michael Hayden, MD, Ph.D, Principal Investigator — University of British Columbia
Locations (1):
- Children's and Women's Health Centre of British Columbia, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Mufti K, Cordova M, Scott EN, Trueman JN, Lovnicki JM, Loucks CM, Rassekh SR, Ross CJD, Carleton BC; Canadian Pharmacogenomics Network for Drug Safety Consortium. Genomic variations associated with risk and protection against vincristine-induced peripheral neuropathy in pediatric cancer patients. NPJ Genom Med. 2024 Nov 5;9(1):56. doi: 10.1038/s41525-024-00443-7. PMID 39500896
- [Derived] Carleton B, Poole R, Smith M, Leeder J, Ghannadan R, Ross C, Phillips M, Hayden M. Adverse drug reaction active surveillance: developing a national network in Canada's children's hospitals. Pharmacoepidemiol Drug Saf. 2009 Aug;18(8):713-21. doi: 10.1002/pds.1772. PMID 19507171
- See also: Related Info — http://www.cpnds.ubc.ca
- See also: Related Info — http://www.genomebc.ca